CLINICAL TRIAL: NCT03198052
Title: CAR-T Targeting GPC3, Mesothelin, Claudin18.2, GUCY2C, B7-H3, PSCA, PSMA, MUC1, TGFβ, HER2, Lewis-Y, AXL, or EGFR for Immunotherapy of Lung Cancer: Phase I Clinical Trial
Brief Title: GPC3/Mesothelin/Claudin18.2/GUCY2C/B7-H3/PSCA/PSMA/MUC1/TGFβ/HER2/Lewis-Y/AXL/EGFR-CAR-T Cells Against Cancers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: Hunan Zhaotai Yongren Medical Innovation Co. Ltd. (Other); Guangdong Zhaotai InVivo Biomedicine Co. Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZZCART-002
Record Dates: First submitted 2017-06-22; First posted 2017-06-23 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Lung Cancer; Cancer; Immunotherapy; CAR-T Cell
Keywords: Lung Cancer; CAR-T Cell Therapy; PSCA; MUC1; HER2; Mesothelin; Lewis-Y; GPC3; AXL; EGFR; B7-H3; Claudin18.2; TGFβ; DAP10; HPK1; PD1; CTLA4; Tigit; Knockdown; SCFV
MeSH Terms: conditions — Lung Neoplasms; Neoplasms | interventions — Mesothelin; Guanylate Cyclase; PSCA protein, human

STUDY DESIGN:
Intervention Model Description: Use engineered CAR-T cells to kill cancer cells with certain targets.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T cell therapy group (Experimental): Patients will receive 3 or more cycles of the CAR-T cells treatment via systemic or regional injection, from 1x10e6/kg-10x10e6/kg weight.
  Interventions: Biological: CAR-T cells targeting GPC3, Mesothelin, Claudin18.2, GUCY2C, B7-H3, PSCA, PSMA, MUC1, TGFβ, HER2, Lewis-Y, AXL, or EGFR

INTERVENTIONS:
Biological: CAR-T cells targeting GPC3, Mesothelin, Claudin18.2, GUCY2C, B7-H3, PSCA, PSMA, MUC1, TGFβ, HER2, Lewis-Y, AXL, or EGFR — CAR-T cells injection: (1-10×10e6/kg CAR-T for each treatment; 3 or more cycles.
  Other Names: Administration of CAR-T cells through vein or interventional technique.

SUMMARY:
The third generation of CAR-T cells that target GPC3, Mesothelin, Claudin18.2, GUCY2C, B7-H3, PSCA, PSMA, MUC1, TGFβ, HER2, Lewis-Y, AXL, or EGFR have been constructed respectively and their anti-cancer function has been verified by multiple in vitro and in vivo studies.Clinical studies will be performed to test the anti-cancer function of the these individual or combination of the CAR-T cells for immunotherapy of human cancer patients with GPC3, Mesothelin, Claudin18.2, GUCY2C, B7-H3, PSCA, PSMA, MUC1, TGFβ, HER2, Lewis-Y, AXL, or EGFR expressions. In this phase I study, the safety, tolerance, and preliminary efficacy of the GPC3/Mesothelin/Claudin18.2/GUCY2C/B7-H3/PSCA/PSMA/MUC1/TGFβ/HER2/Lewis-Y/AXL/EGFR

-CAR-T cell immunotherapy on human cancers will firstly be tested.

DETAILED DESCRIPTION:
1. Choose appropriate patients with advanced lung or other cancers,with written consent for this study;
2. Perform biopsy to determine the expression of HER2, Mesothelin, Lewis-Y, PSCA, MUC1, GPC3, AXL, EGFR, Claudin18.2, or B7-H3 of the tumor by western blotting or IHC;
3. Collect blood from the patients and isolate mononuclear cells, activate the T cells and transfect the T cells with GPC3, Mesothelin, Claudin18.2, GUCY2C, B7-H3, PSCA, PSMA, MUC1, TGFβ, HER2, Lewis-Y, AXL, or EGFR targeting CAR, amplify the transfected T cells as needed, test the quality and killing activity of the CAR-T cells and then transfer them back the patients via systemic or local injections, and follow up closely to collect related results as needed;
4. To enhance the killing capability, CD4+ T cells are genetically engineered to express TGFβ-CAR and secret IL7/CCL19 and/or SCFVs against PD1/CTLA4/Tigit; CD8+T cells are constructed to express GPC3/Mesothelin/Claudin18.2/GUCY2C/B7-H3/PSCA/PSMA/MUC1/TGFβ/HER2/Lewis-Y/AXL/EGFR

   -DAP10-CAR with knockdown of PD1/HPK1;
5. Other cancers with these cell surface antigen expressions are also recruited if needed;
6. Evaluate the clinical results as needed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced cancer that expresses GPC3/Mesothelin/Claudin18.2/GUCY2C/B7-H3/PSCA/PSMA/MUC1/TGFβ/HER2/Lewis-Y/AXL/EGFR protein; 2. Life expectancy >12 weeks; 3. Adequate heart,lung,liver,kidney function; 4. Available autologous transduced T cells with greater than or equal to 20% expression ofGPC3, Mesothelin, Claudin18.2, GUCY2C, B7-H3, PSCA, PSMA, MUC1, TGFβ, HER2, Lewis-Y, AXL, or EGFR-CAR determined by flow-cytometry and killing of GPC3, Mesothelin, Claudin18.2, GUCY2C, B7-H3, PSCA, PSMA, MUC1, TGFβ, HER2, Lewis-Y, AXL, or EGFR-positive targets greater than or equal to 20% in cytotoxicity assay; 5. Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent.

-

Exclusion Criteria:

1. Had accepted gene therapy before;
2. Severe virus infection such as HBV,HCV,HIV,et al;
3. Known HIV positivity;
4. Active infectious disease related to bacteria, virus,fungi,et al;
5. Other severe diseases that the investigators consider not appropriate;
6. Pregnant or lactating women;
7. Systemic steroid treatment (greater than or equal to 0.5 mg prednisone equivalent/kg/day);
8. Other conditions that the investigators consider not appropriate. -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2036-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Dose Limiting Toxicity | three months
  A dose limiting toxicity is defined as any toxicity that is considered to be primarily related to the GPC3/Mesothelin/Claudin18.2/GUCY2C/B7-H3/PSCA/PSMA/MUC1/TGFβ/HER2/Lewis-Y/AXL/EGFR-CAR T cells,which is irreversible, or life threatening or hematologic or non-hematologic Grade 3-5.

SECONDARY OUTCOMES:
Percent of Patients with best response as either complete remission or partial remission. | three months
  Response rates will be estimated as the percent of patients whose best response is either complete remission or partial remission by combining the data from the patients. To compare with historical data, a 95% confidence interval will be calculated for the response rate.
Median CAR-T cell persistence | Six years
  Median CAR-T cell persistence will be measured by quantitative rt-PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenfeng Zhang, MD,PhD, Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University
Locations (2):
- China (2):
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wei X, Lai Y, Li J, Qin L, Xu Y, Zhao R, Li B, Lin S, Wang S, Wu Q, Liang Q, Peng M, Yu F, Li Y, Zhang X, Wu Y, Liu P, Pei D, Yao Y, Li P. PSCA and MUC1 in non-small-cell lung cancer as targets of chimeric antigen receptor T cells. Oncoimmunology. 2017 Feb 6;6(3):e1284722. doi: 10.1080/2162402X.2017.1284722. eCollection 2017. PMID 28405515